CLINICAL TRIAL: NCT06394427
Title: Influence of Neoadjuvant Chemoimmunotherapy on Treatment Response in Stage IIIA- N2IIIB Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Chemoimmunotherapy in Stage IIIA- N2IIIB Non-small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Pengfei Li, Research Assistant, West China Hospital
Other Study IDs: 2024-674
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer Stage ⅢA; Non-small Cell Lung Cancer Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chemoimmunotherapy group 1: patients received different cycles of neoadjuvant chemoimmunotherapy
  Interventions: Other: cycles of neoadjuvant therapy and duration of waiting for surgery
- chemoimmunotherapy group 2: the duration of before patients received surgery after neoadjuvant chemoimmunotherapy
  Interventions: Other: cycles of neoadjuvant therapy and duration of waiting for surgery

INTERVENTIONS:
Other: cycles of neoadjuvant therapy and duration of waiting for surgery — We intended to explore the cycles of neoadjuvant therapy and duration of waiting for surgery on the perioperative outcomes and long-term prognosis of locally advanced NSCLC in the real world

SUMMARY:
to explore the impact of preoperative neoadjuvant immunotherapy on perioperative outcomes and long-term prognosis of locally advanced NSCLC in the real world

ELIGIBILITY:
Inclusion Criteria:

* Confirmed as primary lung cancer through cytology or histological examination;

  * ECOG score of 0 or 1; ③ 18 years old or above;

    * Received imaging examination, with a preliminary clinical staging of stage III;

      * Received genetic testing and tested negative for EGFR mutations, ALK or ROS-1 fusion; ⑥ Accepting preoperative neoadjuvant immunotherapy combined with chemotherapy; ⑦ Receive surgical treatment after completion of neoadjuvant therapy; ⑧ The postoperative specimens were sent to the pathology department of our hospital for pathological testing, and a complete pathological report is available.

Exclusion Criteria:

* Patients with combined small cell lung cancer; ② Patients with severe liver/kidney dysfunction, cardiovascular disease, or systemic immune disorders;

  * Accept other neoadjuvant treatments; ④ Patients participating in any clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced NSCLC meeting the above crateria
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
major pathological remission | one month
  proportion of patients with no more than 10% residual viable tumor cells; patients who showed no viable tumor in the lung primary setting but lymph nodes show viable metastatic carcinoma were also classified as MPR
pathological complete remission | one month
  proportion of patients without residual viable tumor cell on evaluation of resected lung cancer specimens including all sampled regional lymph nodes
survival time | 5 years
  time since diagnosed with NSCLC

IPD SHARING:
Plan to Share IPD: No
The datasets are available upon reasonable request.